CLINICAL TRIAL: NCT00618631
Title: Effects of Smoking on Opioid Receptor Binding Using [(11)C]Carfentanil: An Imaging PET Study
Brief Title: Effects of Smoking on Opioid Receptor Binding: A PET Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Screening
Other Study IDs: 999908060; 08-DA-N060
Record Dates: First submitted 2008-02-17; First posted 2008-02-20 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-01-08

CONDITIONS: Substance-related Discorder
Keywords: Smoking; Nicotine; Endogenous Opioids; PET Study; Carfentanil
MeSH Terms: conditions — Smoking | interventions — Nicotine; carfentanil

INTERVENTIONS:
Drug: Nicotine
Drug: Carfentanil

SUMMARY:
Background:

* Tobacco smoking is one of the most preventable causes of morbidity and mortality in the world, but the addictive property of nicotine is such that fewer than 10 percent of people who attempt to quit smoking remain tobacco-free after 1 year. Researchers are studying the addictive properties of nicotine in an attempt to develop more successful medication therapies for smoking cessation.
* Nicotine acts on chemical receptors in the brain, including opioid receptors that affect the perception of pain. Repeated nicotine administration can cause adaptations in the brain s opioid receptors, which heightens the addictive properties of nicotine and increases the likelihood and severity of withdrawal symptoms associated with smoking cessation. Researchers are interested in using positron emission tomography (PET) scanning to study brain chemical responses to nicotine in current smokers and nonsmokers.

Objectives:

* To study brain chemical activity related to cigarette smoking and nicotine administration.
* To compare the brain chemical activity of current daily smokers with that of nonsmokers.

Eligibility:

- Individuals 21 to 50 years of age who are either current smokers (10 to 25 cigarettes daily for at least 2 years) or have had some exposure to tobacco but have never smoked regularly (may have had a maximum of 20 cigarettes in their lifetime and none in past year).

Design:

* Eligible participants will undergo initial medical and psychological screening and neuropsychological testing before beginning the main phase of the study. Participants will be required to abstain from alcohol and drugs (except caffeine, nicotine, and prescription drugs) for 24 hours before each session, and smokers will refrain from smoking after midnight on the night before each session.
* Session 1: Participants will answer questions about nicotine craving and withdrawal symptoms, followed by a magnetic resonance imaging (MRI) scan to provide baseline information about brain activity.
* Session 2 and 3: Participants will answer questions about nicotine craving and withdrawal symptoms, and then will smoke one cigarette (either active nicotine or placebo). Researchers will document participants consumption of the cigarette. After the cigarette is smoked, participants will have a PET scan. Blood samples will be drawn during the PET session.

DETAILED DESCRIPTION:
Objective: To determine whether nicotine, at the dose delivered through a cigarette (1-2 mg), will increase the release of endogenous opioids, measured by the displacement of the mu-opioid PET receptor radioligand [(11)C]carfentanil and to determine whether smokers have adaptations in the opioid system compared with nonsmokers.

Study Population: 20 current, daily smoikers and 20 never-smokers who have smoked between 1 and 20 cigarettes in their lifetime.

Design: Double-blind, placebo-controlled, parallel groups design.

Outcome Measures: 1) displacement [(11)C]carfentanil binding, secondary to the release of endorphins by nicotine; 2) upregulation of [(11)C]carfentanil specific binding in smokers compared with nonsmokers; 3) [(11)C]carfentanil specific binding as a function of the mu-opioid receptor A118G polymorphism; and 4) correlation between self-report measures of nicotine effect and [(11)C]carfentanil binding profile.

ELIGIBILITY:
* INCLUSION CRITERIA FOR SMOKERS:

  1. 21-50 year old males and females
  2. smoke 10 cigarettes per day on average for at least 2 years
  3. urine cotinine level greater than or equal to 200 ng/ml (NicAlert reading greater than or equal to 4)
  4. estimated IQ score greater than or equal to 85 (competent to give informed consent)
  5. medically and psychologically healthy as determined by screening criteria.

EXCLUSION CRITERIA FOR SMOKERS:

1. interest in reducing or quitting tobacco use
2. treatment for nicotine dependence in the past 3 months
3. current drug or alcohol abuse or dependence
4. consumption of more than 15 alcoholic drinks per week during the past month
5. any opiate use in the past 6 months
6. marijuana use greater than one time per week on an average during the past month
7. other drug use greater than 2 time per month on average during the past 3 months.
8. current use of any medication that would interfere with the protocol
9. under the influence of a drug or alcohol at experimental sessions
10. HIV positive
11. history of psychotropic medications
12. history of head injury with unconscious longer than 5 minutes
13. implantable device or foreign body that would make an MRI examination unobtainable
14. MRI abnormality judged clinically significant by the PI
15. use of any investigational medication or device within the previous 30 days
16. donation at least 450 ml of blood or equivalent levels of plasma within the previous 30 days
17. exposure to ionizing radiation that, in combination with the study tracer, would result in a cumulative exposure exceeding 5 rem in one calendar year
18. any subject judged by the PI to be inappropriate for the study.
19. chronic pulmonary disease, including COPD, bronchitis, asthma, and emphysema
20. pregnant, nursing, or become pregnant during the study

INCLUSION CRITERIA FOR NONSMOKERS:

1. 21-50 year old males and females
2. smoked 1-20 cigarettes in their life and none in past year
3. urine cotinine level less than 30 ng/ml (NicAlert reading less than or equal to 1)
4. estimated IQ score greater than or equal to 85 (competent to give informed consent)
5. medically and psychologically healthy as determined by screening criteria.

EXCLUSION CRITERIA FOR NONSMOKERS:

1. use of any tobacco products in the past year
2. current drug or alcohol abuse or dependence
3. consumption of more than 15 alcoholic drinks per week during the past month
4. any opiate use in the past 6 months
5. marijuana use greater than one time per week on average during past month
6. other drug use greater than two times per month on average during past three months.
7. current use of any medication that would interfere with the protocol
8. under the influence of a drug or alcohol at experimental sessions
9. HIV positive
10. history of psychotropic medications
11. history of head injury with unconscious longer than 5 minutes
12. implantable device or foreign body that would make an MRI examination unobtainable
13. MRI abnormality judged clinically significant by the PI
14. use of any investigational medication or device within the previous 30 days
15. donation of at least 450 ml of blood or equivalent levels of plasma within the previous 30 days
16. exposure to ionizing radiation that, in combination with the study tracer, would result in a cumulative exposure exceeding 5 rem in one calendar year
17. any subject judged by the PI to be inappropriate for the study.
18. chronic pulmonary disease, including COPD, bronchitis, asthma, and emphysema
19. pregnant, nursing, or become pregnant during the study

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-01-17; Study Completion 2015-01-08 (Actual)

PRIMARY OUTCOMES:
Changes in carfentanil binding.

SECONDARY OUTCOMES:
Cardiovascular and subjective responses to smoking one cigarette.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Heishman, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - National Institute on Drug Abuse, Baltimore, Maryland
  - Johns Hopkins Medical Institute, Baltimore, Maryland

REFERENCES:
- [Background] Bencherif B, Guarda AS, Colantuoni C, Ravert HT, Dannals RF, Frost JJ. Regional mu-opioid receptor binding in insular cortex is decreased in bulimia nervosa and correlates inversely with fasting behavior. J Nucl Med. 2005 Aug;46(8):1349-51. PMID 16085593
- [Background] Champtiaux N, Gotti C, Cordero-Erausquin M, David DJ, Przybylski C, Lena C, Clementi F, Moretti M, Rossi FM, Le Novere N, McIntosh JM, Gardier AM, Changeux JP. Subunit composition of functional nicotinic receptors in dopaminergic neurons investigated with knock-out mice. J Neurosci. 2003 Aug 27;23(21):7820-9. doi: 10.1523/JNEUROSCI.23-21-07820.2003. PMID 12944511